CLINICAL TRIAL: NCT01915407
Title: AggreGuide 325 mg. Aspirin Study for Aspirin Induced Platelet Dysfunction
Status: Completed | Type: Observational
Sponsor: Aggredyne, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AGD 051
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Platelet Dysfunction Due to Aspirin Ingestion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To test the AggreGuide A-100 AA Assay's effectiveness for detecting aspirin induced platelet dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* over 18

Exclusion Criteria:

* on aspirin in prior week
* medical history of platelet disorders
* contraindications to aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: aspirin naïve subjects over 18
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Platelet Activity Index (PAI) before and after ingestion of aspirin | 2 - 30 hours post aspirin ingestion
  PAI is the proprietary reporting unit of the Aggreguide. It is related to the amount of platelet aggregation in the sample of whole blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Aggredyne, Inc., Houston, Texas, United States